CLINICAL TRIAL: NCT06988462
Title: Pilot Study of "Bottarga" Supplementation: A Little-known, Sustainable "Blue" Food
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge Health Alliance (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CHA-IRB-24-25-346
Record Dates: First submitted 2025-05-16; First posted 2025-05-23 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Prediabetes
Keywords: Bottarga; pre diabetes; inflammation; sustainability; nutritional intervention; overweight
MeSH Terms: conditions — Prediabetic State; Glucose Intolerance; Inflammation; Overweight

STUDY DESIGN:
Intervention Model Description: A randomized, controlled, open-label, crossover pilot study will investigate the metabolic effects of daily Bottarga supplementation, compared to a calorically matched dairy product, in 20 overweight and pre-diabetic participants. Each intervention will last 8 weeks, separated by a 2-week washout period.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bottarga supplementation (intervention group) (Experimental): Ten overweight and pre-diabetic participants randomly allocated to 8 weeks of daily bottarga supplementation (20 grams/day) as an initial treatment. Baseline assessment measures will be repeated, followed by a 2-week wash-out period. Then, assessment measures will be repeated followed by 8 weeks of daily cream cheese supplementation (28 grams/day), followed by final assessment measures.
  Interventions: Other: Bottarga
- Cream cheese supplementation (control) (Sham Comparator): Ten overweight and pre-diabetic participants randomly allocated to 8 weeks of daily cream cheese supplementation (28 g/day) as the initial intervention. Baseline assessment measures will be repeated, followed by a 2-week wash-out period. Then, assessment measures will be repeated, followed by 8 weeks of daily Bottarga supplementation (20 g/day), followed by final assessment measures.
  Interventions: Other: Comparator

INTERVENTIONS:
Other: Bottarga — Participants will consume prepackaged daily doses of Bottarga, each containing the required amount (20 grams/day) for 8 weeks.
  Arms: Bottarga supplementation (intervention group)
Other: Comparator — Participants will consume 28g of cream cheese/day for 8 weeks.
  Arms: Cream cheese supplementation (control)

SUMMARY:
This pilot study aims to explore the potential benefits of consuming Greek Bottarga (grey mullet fish roe) in overweight, pre-diabetic individuals.

Before initiating the crossover randomized controlled trial (RCT), the investigators will conduct a preliminary dose-testing study in five overweight and pre-diabetic adults.Participants will undergo clinical assessments before and after the dietary intervention to evaluate changes in metabolic health markers. Following this, the investigators will proceed with a randomized, controlled crossover trial involving 20 overweight and pre-diabetic adults. This main study phase will compare the metabolic effects of daily Bottarga supplementation to those of a calorically matched dairy product over an 8-week period, with a 2-week washout period between interventions.

The investigators anticipate that Bottarga supplementation will lead to improvements in lipid profiles, inflammation, and insulin resistance, which could promote the use of sustainable blue foods as part of a healthy diet.

DETAILED DESCRIPTION:
Rationale/goals: Greek Bottarga (Grey mullet fish roe) is a traditional marine or "blue" food "that is produced in a sustainable manner. Bottarga's composition supports that it has excellent nutritional properties, but to date no human/clinical studies have been published. This pilot study will explore the potential benefits of Bottarga consumption in humans. If the results show potential benefits, this would help promote more sustainable blue foods. Methods: Before initiating the crossover randomized controlled trial (RCT), the investigators will conduct a preliminary dose-testing study in five overweight and pre-diabetic adults, who will consume 20 g/day of Bottarga. Participants will undergo clinical assessments before and after the dietary intervention to evaluate changes in metabolic health markers.

The current randomized, controlled, cross-over pilot study (Open Label, Two-Arms) will investigate the metabolic effects of daily bottarga supplementation (versus a calorically equal dairy product) in 20 overweight and pre-diabetic participants for 8 weeks with a 2-week "washout" period between food supplement arms. The primary outcome will be determined based on the most clinically important results observed during phase 1. Anticipated Results: The investigators expect Bottarga supplementation to be associated with more beneficial changes on lipid profiles, inflammatory markers and insulin resistance compared to baseline measures and to the calorically equivalent comparator food.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 60 years
* Residents of Massachusetts
* Diagnosed with prediabetes
* Body Mass Index (BMI) greater than 27 kg/m²
* Otherwise healthy
* Not pregnant
* Willing to take a nutritional supplement

Exclusion Criteria:

* Use of any medications for diabetes, dyslipidemia, or immunosuppression
* Current use of any supplements containing n-3 fatty acids
* Current use of tobacco/nicotine products, marijuana, or illicit drugs
* Self-reported consumption of a diet rich in plant- or marine-derived fats (e.g., fatty fish, nuts, seeds, or olive oil)
* Use of hormone therapy (except oral contraceptives)
* Known allergies to fish, seafood, or any fish-derived products, including bottarga
* Pregnancy
* Clinical evidence or history of cardiac, pulmonary, hepatic, or renal insufficiency
* Immunodeficiency conditions
* History of non-skin cancer
* Participation in other clinical research studies

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-25 (Estimated); Primary Completion 2025-11-25 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Mean change in fasting glucose | From baseline (start of the intervention) to Week 8 (end of the initial intervention period, prior to crossover), and from Week 10 to Week 18 (end of the second intervention period following crossover).
  Mean change in fasting glucose levels (mg/dL) after overnight fast.
Mean Change in High-Sensitivity C-Reactive Protein (hs-CRP) | From baseline (start of the intervention) to Week 8 (end of the initial intervention period, prior to crossover), and from Week 10 to Week 18 (end of the second intervention period following crossover).
  Mean change in serum hs-CRP levels (mg/L) after overnight fast.
Mean Change in Hemoglobin A1c (HbA1c) | From baseline (start of the intervention) to Week 8 (end of the initial intervention period, prior to crossover), and from Week 10 to Week 18 (end of the second intervention period following crossover).
  Mean change in HbA1c levels (%) after overnight fast.
Mean Change in Lipid Profile (Total Cholesterol, Triglycerides, HDL-C, LDL-C) | From baseline (start of the intervention) to Week 8 (end of the initial intervention period, prior to crossover), and from Week 10 to Week 18 (end of the second intervention period following crossover).
  Mean change in fasting lipid levels-including total cholesterol (mg/dL), triglycerides (mg/dL), high-density lipoprotein cholesterol (HDL-C, mg/dL), and low-density lipoprotein cholesterol (LDL-C, mg/dL after overnight fast.

SECONDARY OUTCOMES:
Mean change in body mass index | From baseline (start of the intervention) to Week 8 (end of the initial intervention period, prior to crossover), and from Week 10 to Week 18 (end of the second intervention period following crossover).
  Body Mass Index (kg/m-squared)
Mean change in body fat | From baseline (start of the intervention) to Week 8 (end of the initial intervention period, prior to crossover), and from Week 10 to Week 18 (end of the second intervention period following crossover).
  Body fat percentage as measured by bioelectrical impedance
Mean change in waist circumference | From baseline (start of the intervention) to Week 8 (end of the initial intervention period, prior to crossover), and from Week 10 to Week 18 (end of the second intervention period following crossover).
  Waist circumference (cm)
Mean change in waist/hip ratio | From baseline (start of the intervention) to Week 8 (end of the initial intervention period, prior to crossover), and from Week 10 to Week 18 (end of the second intervention period following crossover).
  Waist/hip ratio (waist circumference (cm) divided by hip circumference (cm)
Mean change in resting blood pressure | From baseline (start of the intervention) to Week 8 (end of the initial intervention period, prior to crossover), and from Week 10 to Week 18 (end of the second intervention period following crossover).
  Resting systolic and diastolic blood pressure (mmHg), measured using calibrated automated sphygmomanometers.
Mean change in liver enzymes | From baseline (start of the intervention) to Week 8 (end of the initial intervention period, prior to crossover), and from Week 10 to Week 18 (end of the second intervention period following crossover).
  Aspartate aminotransferase (AST, U/L), Alanine aminotransferase (ALT, U/L), Alkaline phosphatase (ALP, U/L) after overnight fast.

CONTACTS AND LOCATIONS:
Overall Officials: Stefanos N Kales, Professor of Medicine, Harvard Medical School, MD, Principal Investigator — Cambridge Health Alliance
Locations (1):
- Cambridge Health Alliance, Sommerville, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided